CLINICAL TRIAL: NCT01173549
Title: A Double-Blind, Randomized, Placebo Controlled, 2-Period Crossover Study to Evaluate the Effect of a Single Dose of JNJ-28431754 (Canagliflozin) on Gastrointestinal Glucose Absorption and Metabolism in Healthy Subjects
Brief Title: A Study of 28431754 (Canagliflozin) on Gastrointestinal Glucose Absorption and Metabolism in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Study Physician, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CR017224; 28431754DIA1022
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Canagliflozin; Pharmacodynamic; Glucose absorption; Glucose metabolism
MeSH Terms: interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 001 (Experimental): no intervention Part 1: 240 mL water 10 minutes (min) prior to the start of the MMTT on Day 1 of Periods 1 and 2. Periods 1 and 2 will be separated by 7 to 21 days.
  Interventions: Other: no intervention
- 002 (Experimental): Canagliflozin/Placebo Placebo/Canagliflozin Part 2: 240 mL water 20 min prior to the MMTT on Day 1 of Periods 1 and 2 in each treatment sequence (1 dose of canagliflozin in Period 1 followed by 1 dose of placebo in Period 2 and then crossover to 1 dose of placebo in Period 1 followed by 1 dose of canagliflozin in Period 2).
  Interventions: Drug: Canagliflozin/Placebo Placebo/Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin/Placebo Placebo/Canagliflozin — Part 2: 240 mL water 20 min prior to the MMTT on Day 1 of Periods 1 and 2 in each treatment sequence (1 dose of canagliflozin in Period 1 followed by 1 dose of placebo in Period 2 and then crossover to 1 dose of placebo in Period 1 followed by 1 dose of canagliflozin in Period 2).
  Arms: 002
Other: no intervention — Part 1: 240 mL water 10 minutes (min) prior to the start of the MMTT on Day 1 of Periods 1 and 2. Periods 1 and 2 will be separated by 7 to 21 days.
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the effect of canagliflozin on gastrointestinal glucose absorption in healthy volunteers.

DETAILED DESCRIPTION:
This is a single center study that will be conducted in two Parts (Part 1 and Part 2) to evaluate the effect of a single-dose of canagliflozin on the absorption of glucose in healthy volunteers. Part 1 is a pilot (small) study where responses to key pharmocodynamic (PD) parameters (ie, specific tests on blood samples to evaluate effects of no treatment on the body) will be measured to confirm the study design and number of volunteers planned for Part 2. Part 2 is the main study where volunteers will be randomized (assigned to study drug or placebo by chance) to receive double-blind (neither the volunteer or study physician will know the identity of the treatment assigned) treatment with canagliflozin or placebo (treatment identical in appearance to canagliflozin but contains no active drug) to evaluate the effect of canagliflozin compared to placebo on gastrointestinal glucose absorption using a radiolabeled glucose tracer approach (ie, where a radioactive substance is combined with glucose allowing the movement of glucose in the body to be traced or detected). Blood and urine samples will be collected from volunteers at pre-defined times during the study for PD analysis. Safety will be monitored during the study by evaluating adverse events and results from clinical laboratory tests, vital signs measurements, electrocardiograms (ECGs), and physical examinations performed. Volunteers in Part 1 will receive 240 ml of water 10 minutes before starting of the MMTT in each period (Periods 1 and 2). Volunteers in Part 2 will receive study drug 20 minutes prior to starting of the MMTT in treatment sequence 1 (a single 300-mg dose of canagliflozin in Period 1 followed by matching placebo in Period 2) or in treatment Sequence 2 (matching placebo in Period 1 followed by a single 300-mg dose of canagliflozin in Period 2). Periods 1 and 2 will be separated by 7 to 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) between 20 and 27 kg/m2 (inclusive) and a body weight not less than 50 kg
* Be healthy on the basis of physical examination including medical history, vital signs, 12-lead ECG, and all other screening lab tests performed at Screening and Admission
* Agree (if men) to use a double barrier method of birth control (e.g., condom for them and use of spermacide with diaphragm, hormonal contraceptives or intrauterine devices by female partner) during the study and for three months following the last dose of study medication, and to not donate sperm during the study and for 3 months after receiving the last dose of study medication
* Willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Must have signed an informed consent form.

Exclusion Criteria:

* Have a history of, or currently active, illness or medical condition or disorder that the Investigator considers to be clinically significant
* Has been a smoker or tobacco user within the past 6 months
* Have a history of recent major surgery (within 6 months of study start)
* Tested positive for serology: hepatitis B surface antigen (HBsAg), hepatitis C antibodies (anti-HCV) or human immunodeficiency virus (HIV) antibodies
* Fasting plasma glucose > 110 mg/dL
* Have a history of alcohol or drug abuse within 2 years prior to Screening or a positive test for alcohol and/or drugs of abuse (including but not limited to barbiturates, opiates, cocaine, cannabinoids, amphetamines,MDMA (Ecstasy) and benzodiazepines) at Screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11; Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The amount of ingested glucose that is absorbed in systemic circulation | During the first 1 and 2 hours after a standard mixed meal

SECONDARY OUTCOMES:
The amount of ingested glucose that is absorbed in systemic circulation | 2-6 hr and 0-6 hr after a standard mixed meal
Endogenous glucose production (EGP) | At protocol-specified time points after a standard mixed meal
Total and incremental plasma glucose and insulin area under the curve (AUC) | 0-1, 0-2, 2-6, and 0-6 hours after a standard mixed meal
Gastric emptying: peak level, time to peak level, and AUCs | 0-6 hours after a standard mixed meal
Rate of Peripheral glucose disposal (Rd) | At protocol-specified time points after a standard mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- La Jolla, California, United States

REFERENCES:
- [Derived] Polidori D, Sha S, Mudaliar S, Ciaraldi TP, Ghosh A, Vaccaro N, Farrell K, Rothenberg P, Henry RR. Canagliflozin lowers postprandial glucose and insulin by delaying intestinal glucose absorption in addition to increasing urinary glucose excretion: results of a randomized, placebo-controlled study. Diabetes Care. 2013 Aug;36(8):2154-61. doi: 10.2337/dc12-2391. Epub 2013 Feb 14. PMID 23412078